CLINICAL TRIAL: NCT01842022
Title: The Effect of the Glycemic Load of Meals on the Cognition and Mood of Older Adults With Differences in Glucose Tolerance
Brief Title: The Effect of the Glycemic Load of Meals on the Cognition and Mood of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, David Benton, Professor of Psychology, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DB-0413
Record Dates: First submitted 2013-04-09; First posted 2013-04-29 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Dementia
Keywords: Glycemic load; memory; mood
MeSH Terms: conditions — Dementia | interventions — isomaltulose; Sucrose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Better glucose tolerance (Other): Take meals with isomaltulose, sucrose or glucose
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose; Dietary Supplement: Glucose
- Better glucose tolerance / Levels fall (Other): Take meals with isomaltulose, sucrose or glucose
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose; Dietary Supplement: Glucose
- Poorer tolerance levels remain high (Other): Take meals with isomaltulose, sucrose or glucose
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose; Dietary Supplement: Glucose
- Poorer glucose tolerance / Levels fall (Other): Take meals with isomaltulose, sucrose or glucose
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose; Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Isomaltulose — Isomaltulose sweetened meal will be given to each of four groups who differ in their glucose tolerance
Dietary Supplement: Sucrose — Sucrose sweetened meal will be given to each of four groups who differ in their glucose tolerance
Dietary Supplement: Glucose — Glucose sweetened meal will be given to each of four groups who differ in their glucose tolerance

SUMMARY:
A lower rather than a higher glycemic load (GL) meal has been shown to benefit cognition and mood, however, the data in older adults and those most prone to cognitive dysfunction, is limited and conflicting. One explanation is that the GL of a meal may interact with a person's pre-existing glucose tolerance (GT).

As older adults have a higher incidence of glucose tolerance and are more likely to experience memory problems the present study considers the interaction between the GL of meal in those with better or poorer GT.

The population studied will not have a history of diabetes or dementia. A battery of cognitive tests will be administered after meals sweetened with one of three sugars known to vary in the rate that they release glucose into the blood stream.

DETAILED DESCRIPTION:
On day one subjects will take an oral glucose tolerance test and will then be divided into four groups depending on their glucose tolerance (how long values remain raised) and the tendency for values to subsequently fall to low values.

On a second occasion 155 healthy older adults, aged 45-80 years, will be randomly assigned to receive either a glucose, sucrose or isomaltulose based meal. All meals are matched on macronutrient composition and differ only in glycemic load. Cognitive performance and mood will be assessed 30, 105 and 180 minutes after breakfast. Measures of memory, attention, reaction times and mood will be taken.

The response to the three meals will be contrasted in those with different glucose profiles on day one

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of 45 to 80 years

Exclusion Criteria:

* Type 1 or type 2 diabetes
* Dementia
* Liver disease
* Gastro-intestinal problems

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in episodic memory | 30, 105, 180 minutes
  Episodic memory assessed by asking subjects to recall a list of words

SECONDARY OUTCOMES:
Change in mood | 30, 105, 180 minutes
  Visual analogues scales used to report mood at six points during study

OTHER OUTCOMES:
Change in reaction Times | 30, 105, 180 minutes
  1,2,4 and 8 lamps will be monitored and the time taken to extinguish will be measured
Change in vigilance | 30, 105 and 180 minutes
  Digits will be generated at rate of 100 per minute. Subjects indicate when they see either three odd or three even in a row

CONTACTS AND LOCATIONS:
Overall Officials: David Benton, DSc, Principal Investigator — Swansea University
Locations (1):
- Psychology, Swansea University, Swansea, Wales, United Kingdom